CLINICAL TRIAL: NCT05033236
Title: Platelets and Complement Activation in Coronary Artery Bypass Graft Surgery (CABG)
Acronym: PAC
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1097/2018
Record Dates: First submitted 2020-06-10; First posted 2021-09-02 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Cardiopulmonary Bypass; Inflammatory Response; Platelet Dysfunction
Keywords: bleeding; transfusion; cardiopulmonary bypass; cardiac surgery; complement system
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients undergoing coronary artery bypass graft surgery (CABG) frequently exhibit postoperative bleeding complications which are still a major cause for morbidity and mortality. One major contributing factor is the loss of platelets and impaired platelet function. During cardiopulmonary bypass (CPB) blood comes in close contact with foreign surfaces which induces a series of reactions; especially the complement system as part of the innate immunity is highly activated. Due to the strong crosslink between complement system, platelet function and the plasmatic coagulation it is likely that complement activation during CPB has an impact on the overall process of clot formation. Besides the activation of the complement system there is growing evidence that the occurrence of mitochondrial DNA (mtDNA) during CPB might be related to further platelet activation . Activated platelets may enhance micro-thrombosis leading to organ failure and thereby contributing to postoperative morbidity.

One major complication during and after CABG surgery is bleeding requiring transfusion and even reoperation in about 2%- 8% of patients.

As bleeding complications increase patient morbidity and mortality, this study is designed to investigate the possible mechanisms of platelet loss during CABG.

The hypothesis is that increased complement activation during CPB leads to platelet activation and loss of platelets. Further the degree of complement activation and levels of mtDNA might correlate with postoperative bleeding, transfusion requirements and clinical outcome.

DETAILED DESCRIPTION:
2.1. Primary Study Objective The aim of the study is to examine the correlation between complement activation (c5b-9) and platelet decline during elective coronary artery bypass graft (CABG) on cardiopulmonary bypass (CPB).

2.2. Further Study Objectives A secondary aim of the study is to investigate the specific pathway of complement activation, the mtDNA levels and the interaction with platelet function.

Therefore correlations between levels of complement factors [c5b-9, C1q (C1r/C1s), C3a, C5a, MBL, Factor B, Factor D], mtDNA level [human NADH dehydrogenase 1 gene] and platelet function [MPV/PTC ratio and FACS for platelet activation factor 4 (PFA)] will be examined.

Further it will be explored whether the level of complement activation and levels of mtDNA and the plasmatic coagulation system correlate with transfusion requirements, postoperative morbidity (need for revision surgery, cardiovascular events including thromboembolic events, sepsis, single or multiple organ failure according to SOFA Score), and in hospital mortality.

There will be also a correlation conducted between levels of complement [see above] and concentration of coagulation factors [F I - F XIII, FXa, FXIIa, Kallikrein, Bradykinin, endogenous thrombin potential (ETP)], transfusion requirements, mtDNA and platelet function to postoperative morbidity (need for revision surgery, cardiovascular events including thromboembolic events, sepsis, single or multiple organ failure according to SOFA Score) and in hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

I.1. Male and female subjects > 18 years and < 86 years I.2. elective coronary artery bypass graft surgery with or without valve surgery (max. 2 valves) and elective valve surgery (max. 2 valves) on cardiopulmonary bypass (CPB) I.3. ASA I - IV I.4. written informed consent

Exclusion Criteria:

E.1. emergency CABG with or without cardiac valve surgery and emergency valve surgery and emergency aortic dissection E.2. preexisting complement deficiency syndromes E.3. preexisting thrombocytopathy or thrombocytopenia (platelet count below 100 G/L) E.4. Known history of congenital coagulopathy E.5. Patients that are known to be pregnant E.6 Known participation in another interventional clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation
Study Population: elective cardiac surgery patients scheduled for CPB procedure meeting the inclusion criteria at the University Hospital Innsbruck
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
correlation between complement activation (c5b-9) and platelet decline | 4 days
  The aim of the study is to examine the correlation between complement activation (c5b-9) and platelet decline during elective coronary artery bypass graft (CABG) with or without valve surgery (max. 2 valves) and elective valve surgery (max. 2 valves) on cardiopulmonary bypass (CPB).

SECONDARY OUTCOMES:
A secondary aim of the study is to investigate the specific pathway of complement activation, the mtDNA levels and the interaction with platelet function. | 4 days
  Therefore we search for correlations between levels of complement factors [c5b-9, C1q (C1r/C1s), C3a, C5a, MBL, Factor B, Factor D], mtDNA level [human NADH dehydrogenase 1 gene] and platelet function [MPV/PTC ratio and FACS for platelet activation factor 4 (PFA)].

CONTACTS AND LOCATIONS:
Overall Officials: Judith Martini, MD, Prof., Principal Investigator — Medical University Innsbruck - Anesthesia and Intensive Care
Locations (1):
- University Hospital Innsbruck, Innsbruck, Tyrol, Austria

DOCUMENTS (2):
  • Study Protocol (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT05033236/Prot_000.pdf
  • Informed Consent Form (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT05033236/ICF_001.pdf